CLINICAL TRIAL: NCT03583372
Title: An International Phase 3, Randomized, Double-Blind, Active (Tolterodine)-Controlled Multicenter Extension Study to Evaluate the Long-Term Safety and Efficacy of Vibegron in Patients With Symptoms of Overactive Bladder
Brief Title: An Extension Study to Examine the Safety and Tolerability of a New Drug in Patients With Symptoms of Overactive Bladder (OAB).
Acronym: Empowur
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Urovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-901-3004; 2017-003294-33 (EudraCT Number)
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Results first posted 2021-02-03 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Overactive Bladder
Keywords: Beta-3 adrenergic receptor (β3-AR) agonists; incontinence; OAB; vibegron; urge urinary incontinence; Urinary bladder, overactive; Urologic Diseases; Lower Urinary Tract Symptoms; Urological Agents
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urologic Diseases; Lower Urinary Tract Symptoms | interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vibegron + Placebo to match Tolterodine (Experimental)
  Interventions: Drug: Vibegron; Drug: placebos
- Tolterodine + Placebo to match vibegron (Active Comparator)
  Interventions: Drug: placebos; Drug: Tolterodine Tartrate ER

INTERVENTIONS:
Drug: Vibegron — single daily dose 75 mg
  Other Names: RVT-901, MK-4618, KRP114V
  Arms: Vibegron + Placebo to match Tolterodine
Drug: placebos — placebo to match vibegron (experimental drug) and tolterodine (active comparator)
Drug: Tolterodine Tartrate ER — single daily dose of 4 mg
  Other Names: Mariosea XL
  Arms: Tolterodine + Placebo to match vibegron

SUMMARY:
This study is designed to evaluate the safety, tolerability, and efficacy of vibegron administered once daily in participants with OAB for up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Has completed participation in study RVT-901-3003.
2. Has demonstrated ≥ 80% compliance with self-administration of Study Treatment in study RVT-901-3003.

Exclusion Criteria:

1. Has a change in history or current evidence of any clinically significant condition, therapy, lab abnormality, or other circumstance that might, in the opinion of the Investigator, confound the results of the study, interfere with the participant's ability to comply with study procedures, or make participation in the study not in the participant's best interest.
2. Has coronary or neurovascular interventions planned during the duration of the study.
3. Has uncontrolled hyperglycemia (defined as fasting blood glucose >150 mg/dL or 8.33 mmol/L and/or non-fasting blood glucose >200 mg/dL or 11.1 mmol/L) based on most recent available lab results in study RVT-901-3003 or, if in the opinion of the Investigator, is uncontrolled.
4. Has uncontrolled hypertension (systolic blood pressure of ≥ 180 mm Hg and/or diastolic blood pressure of ≥ 100 mm Hg) or has a resting heart rate (by pulse) > 100 beats per minute.
5. Has clinically significant ECG abnormality which, in the opinion of the Investigator, exposes the participant to risk by participating in the study
6. Has alanine aminotransferase or aspartate aminotransferase > 2.0 times the upper limit of normal (ULN), or bilirubin (total bilirubin) > 1.5 x ULN (or > 2.0 x ULN if secondary to Gilbert syndrome or pattern consistent with Gilbert syndrome) based on most recent available lab results in study RVT-901-3003.
7. Has an estimated glomerular filtration rate (eGFR) < 30mL/min/1.73 m2 based on most recent available lab results in study RVT-901-3003.
8. Use of any prohibited medications as detailed in Section 7.7.3.
9. Plans to initiate or change the dosing of any medications listed in Section 7.7.5 during the study that in the opinion of the investigator is assessed to be clinical significant.
10. Has an allergy, intolerance, or a history of a significant clinical or laboratory adverse experience associated with any of the active or inactive components of the vibegron formulation or tolterodine formulation.
11. Is currently participating or has participated in a study with an investigational compound or device within 28 days of signing informed consent, not including participation in study RVT-901-3003.
12. Has a history of significant drug or alcohol abuse/dependence within a year of informed consent, as assessed by the investigator.
13. Has a varying sleep schedule anticipated during times when the voiding diaries are to be completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (107):
- United States (107):
  - Coastal Clinical Research Inc., Mobile, Alabama
  - Clinical Research Consortium, Tempe, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - Core Healthcare Group, Cerritos, California
  - American Clinical Trials, Hawaiian Gardens, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - Prime-Care Clinical Research, Laguna Hills, California
  - Long Beach Clinical Trials LLC, Long Beach, California
  - Downtown L.A. Research Center Inc., Los Angeles, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - Northern California Research, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - WR MCCCR, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Bayview Research Group LLC, Valley Village, California
  - Horizons Clinical Research Center, Denver, Colorado
  - Lynn Institute of Denver, Denver, Colorado
  - Clinical Research Consulting LLC, Milford, Connecticut
  - Coastal Connecticut Research LLC, New London, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - PAB Clinical Research, Brandon, Florida
  - Top Medical Research Inc., Cutler Bay, Florida
  - Revival Research, Doral, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Indago Research Health Center, Hialeah, Florida
  - Best Quality Research, Inc., Hialeah, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - San Marcus Research Clinic Inc., Miami, Florida
  - LCC Medical Research Institute Inc., Miami, Florida
  - Nuren Medical Research Center, Miami, Florida
  - AppleMed Research Group LLC, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Advanced Medical Research Institute, Miami, Florida
  - Suncoast Clinical Research Inc., New Port Richey, Florida
  - Bayside Clinical Research, New Port Richey, Florida
  - Compass Research LLC, Orlando, Florida
  - South Broward Research LLC, Pembroke Pines, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - In-Quest Medical Research, LLC, Peachtree Corners, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Evanston Premier Healthcare Research, Evanston, Illinois
  - Clinical Investigation Specialists Inc., Gurnee, Illinois
  - Investigators Research Group LLC, Brownsburg, Indiana
  - Central Kentucky Research Associates Inc., Lexington, Kentucky
  - DelRicht Research, New Orleans, Louisiana
  - Regional Urology LLC, Shreveport, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Infinity Medical Research Inc., North Dartmouth, Massachusetts
  - Bay State Clinical Trials Inc., Watertown, Massachusetts
  - Remidica LLC, Rochester, Michigan
  - Montana Health Research Institute Inc., Billings, Montana
  - Barrett Clinic P.C., La Vista, Nebraska
  - Women's Clinic of Lincoln PC, Lincoln, Nebraska
  - Meridian Clinical Research LLC, Norfolk, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - Premier Urology Group LLC, Edison, New Jersey
  - Urologic Research and Consulting LLC, Englewood, New Jersey
  - Lawrence OB-GYN Clinical Research LLC, Lawrenceville, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - AccumetRx Clinical Research - Division of Urology Group of New Mexico, Albuquerque, New Mexico
  - United Medical Associates, Binghamton, New York
  - Regional Clinical Research Inc., Endwell, New York
  - AccuMed Research Associates, Garden City, New York
  - Drug Trials America, Hartsdale, New York
  - Upstate Clinical Research Associates LLC, Williamsville, New York
  - PMG Research of Charlotte LLC, Charlotte, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - PMG Research, Wilmington, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Sentral Clinical Research Services, Cincinnati, Ohio
  - Rapid Medical Research, Cleveland, Ohio
  - Buckeye Health and Research, Columbus, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - Providence Health Partners, Dayton, Ohio
  - HWC Womens Research Center, Englewood, Ohio
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - Family Practice Center of Wadsworth Inc. - New Venture Medical Research, Wadsworth, Ohio
  - Ohio Clinical Research LLC, Willoughby Hills, Ohio
  - Leonard Maliver MD Antria, Inc., Indiana, Pennsylvania
  - The Clinical Trial Center LLC, Jenkintown, Pennsylvania
  - Clinical Research of Philadelphia LLC, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians Inc., Pittsburgh, Pennsylvania
  - Research Protocol Management Specialists Hills ObGyn Associates Inc, Pittsburgh, Pennsylvania
  - Greater Providence Clinical Research, LLC, East Providence, Rhode Island
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Piedmont Research Partners, Fort Mill, South Carolina
  - Family Medicine of SayeBrook LLC, Myrtle Beach, South Carolina
  - Hillcrest Clinical Research LLC, Simpsonville, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - MultiSpecialty Clinical Research, Inc., Johnson City, Tennessee
  - Adams Patterson Gynecology and Obstetrics, Memphis, Tennessee
  - DiscoveResearch Inc., Bryan, Texas
  - WR Global Medical Research, DeSoto, Texas
  - Advances in Health, Houston, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - Clinical Trials of Texas Inc., San Antonio, Texas
  - Bandera Family Health Care, San Antonio, Texas
  - Wasatch Clinical Research LLC, Salt Lake City, Utah
  - Health Research of Hampton Roads Inc., Newport News, Virginia
  - Seattle Urology Research, Burien, Washington
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Staskin D, Frankel J, Varano S, Shortino D, Jankowich R, Mudd PN Jr. Once-Daily Vibegron 75 mg for Overactive Bladder: Long-Term Safety and Efficacy from a Double-Blind Extension Study of the International Phase 3 Trial (EMPOWUR). J Urol. 2021 May;205(5):1421-1429. doi: 10.1097/JU.0000000000001574. Epub 2020 Dec 28. PMID 33356445

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 506 participants with overactive bladder (OAB) who completed 12 weeks in Study RVT-901-3003 (NCT03492281) and were screened and randomized for this extension study, 505 received at least 1 dose of double-blind study drug (Safety Set Extension [SAF-Ext]: vibegron, N = 273; tolterodine, N = 232).
Groups:
- 40 Weeks Vibegron 75 mg: Participants who had been randomized to the placebo group in Study RVT-901-3003 were randomized to receive blinded study treatment of vibegron 75 mg once daily for 40 weeks. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
- 52 Weeks Vibegron 75 mg: Participants who had been randomized in Study RVT-901-3003 to receive vibegron 75 milligrams (mg) were to continue their same treatment once daily in a blinded fashion for 40 weeks. Thus, through participation in both Study RVT-901-3003 and this extension study, participants originally randomized to vibegron 75 mg were to receive 52 weeks total of vibegron. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
- 40 Weeks Tolterodine ER 4 mg: Participants who had been randomized to the placebo group in Study RVT-901-3003 were randomized to receive blinded study treatment of tolterodine extended release (ER) 4 mg once daily for 40 weeks. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
- 52 Weeks Tolterodine ER 4 mg: Participants who had been randomized in Study RVT-901-3003 to receive tolterodine ER 4 mg were to continue their same treatment once daily in a blinded fashion for 40 weeks. Thus, through participation in both Study RVT-901-3003 and this extension study, participants originally randomized to tolterodine ER 4 mg were to receive 52 weeks total of tolterodine ER. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
Period: Overall Study
Arm/Group | 40 Weeks Vibegron 75 mg | 52 Weeks Vibegron 75 mg | 40 Weeks Tolterodine ER 4 mg | 52 Weeks Tolterodine ER 4 mg
Started | 92 | 182 | 91 | 141
Completed | 79 | 156 | 72 | 123
Not Completed | 13 | 26 | 19 | 18
Not completed — Withdrawal by Subject | 6 | 11 | 7 | 8
Not completed — Lost to Follow-up | 4 | 6 | 3 | 2
Not completed — Adverse Event | 1 | 3 | 4 | 4
Not completed — Physician Decision | 0 | 1 | 1 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Subject Withdrawn due to Sponsor | 0 | 0 | 0 | 1
Not completed — Did Not Receive Study Drug | 0 | 1 | 0 | 0
Not completed — Captured as Other in the Database | 1 | 2 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for all participants who received at least 1 dose of study treatment during this extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | 40 Weeks Vibegron 75 mg | 52 Weeks Vibegron 75 mg | 40 Weeks Tolterodine ER 4 mg | 52 Weeks Tolterodine ER 4 mg | Total
Number analyzed (Participants) | 92 | 181 | 91 | 141 | 505
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (13.69) | 62.1 (12.39) | 62.1 (12.14) | 60.6 (12.98) | 61.1 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 140 | 70 | 112 | 395
  Male | 19 | 41 | 21 | 29 | 110
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 2
  Asian | 4 | 16 | 8 | 11 | 39
  Black or African American | 14 | 23 | 10 | 26 | 73
  White | 72 | 141 | 72 | 102 | 387
  Other | 0 | 1 | 1 | 2 | 4
Overactive Bladder (OAB) Type [Count of Participants; unit: Participants] — Urgency incontinence is the involuntary loss of urine accompanied by urgency (referred to as OAB Wet). In the absence of incontinence, OAB is referred to as OAB Dry.
  Participants
    Wet | 71 | 146 | 70 | 108 | 395
    Dry | 21 | 35 | 21 | 33 | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Type of Treatment-emergent Adverse Event
Description: Adverse events were collected in participants with overactive bladder (OAB) who previously completed treatment in Study RVT-901-3003. The treatment-emergent period was defined as the period of time from the first dose date of the active double-blind study treatment, whether in Study RVT-901-3003 or Study RVT-901-3004, through 28 days after the last dose of study treatment, or the date of initiation of another investigational agent or surgical intervention, whichever occurred first.
Time Frame: up to 56 weeks
Population: Safety Extension Set (SAF-Ext) Population: all participants who received at least 1 dose of double-blind study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received. Adverse event datasets for Study RVT-901-3003 and Study RVT-901-3004 were combined for the safety analyses.
Measure: Number; unit: participants
Groups:
- Overall Vibegron 75 mg: Participants who received 40 weeks and 52 weeks vibegron 75 milligrams (mg). Participants who had been randomized to the placebo group in Study RVT-901-3003 were randomized to receive blinded study treatment of vibegron 75 mg once daily for 40 weeks in RVT-901-3004. Participants who received 52 weeks vibegron 75 mg were randomized to receive vibegron 75 mg in both studies. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
- Overall Tolterodine ER 4 mg: Participants who received 40 weeks and 52 weeks tolterodine ER 4 mg. Participants who had been randomized to the placebo group in RVT-901-3003 were randomized to receive blinded study treatment of tolterodine ER 4 mg once daily for 40 weeks in Study RVT-901-3004. Participants who received 52 weeks tolterodine ER 4 mg were randomized to receive tolterodine ER 4 mg in both studies. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
Arm/Group | Overall Vibegron 75 mg | Overall Tolterodine ER 4 mg
Number analyzed (Participants) | 273 | 232
participants
  Any TEAE | 171 | 126
  Any study drug-related TEAE | 59 | 46
  Any Grade ≥ 3 TEAE | 10 | 8
  Any Grade ≥ 3 study drug-related TEAE | 1 | 1
  Any treatment-emergent (TE) SAE | 9 | 10
  Any study drug-related TE SAE | 1 | 2
  Any TEAE leading to discontinuation of study drug | 4 | 8
  Any TEAE of clinical interest | 41 | 32
  Any study drug-related TEAE of clinical interest | 14 | 10

2. Secondary Outcome: Change From Baseline (CFB) at Week 52 in the Average Number of Micturitions Per 24 Hours in All Overactive Bladder (OAB) Participants
Description: A micturition/void is defined as "Urinated in Toilet" as indicated on the Patient Voiding Diary (PVD). The number of micturitions is defined as the number of times a participant voided in the toilet as indicated in the PVD. The average daily number of micturitions was calculated using the daily entries in the PVD (which was to be completed prior to each study visit) as the total number of micturitions that occurred on a Complete Diary Day (CDD) divided by the number of CDDs in the PVD. CFB was calculated as the post-BL value minus the BL value. "Per 24 hours" corresponds to one Diary Day (i.e., time between when the participant got up for the day each morning and time the participant got up for the day the next morning as recorded in the PVD). Covariates included in the mixed model for repeated measures (MMRM) were study visit, treatment, treatment by study visit interaction, Baseline, and the statistically significant terms in Study RVT-901-3003: OAB type (Wet versus Dry) and sex.
Time Frame: Baseline; Week 52
Population: Full Analysis Set Extension (FAS-Ext) Population: all randomized OAB participants who took at least 1 dose of double-blind study treatment during this extension study and had at least 1 subsequent evaluable CFB micturition measurement in this extension study. Only participants with evaluable data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: micturitions per 24 hours
Arm/Group | 52 Weeks Vibegron 75 mg | 52 Weeks Tolterodine ER 4 mg
Number analyzed (Participants) | 152 | 120
micturitions per 24 hours | -2.4 (0.24) | -2.0 (0.26)
Statistical Analysis 1: Comparison: 52 Weeks Vibegron 75 mg; Test type: Other — Estimation of within treatment group change from Baseline; Least squares mean = -2.4, 95% CI 2-sided [-2.9 to -2.0]
Statistical Analysis 2: Comparison: 52 Weeks Tolterodine ER 4 mg; Test type: Other — Estimation of within treatment group change from Baseline; Least squares mean = -2.0, 95% CI 2-sided [-2.5 to -1.5]

3. Secondary Outcome: CFB at Week 52 in the Average Number of Urge Urinary Incontinence (UUI) Episodes Per 24 Hours in OAB Wet Participants
Description: The number of UUI episodes is defined as the number of times a participant had checked "urge" as the main reason for the leakage in the PVD, regardless of whether more than one reason for leakage in addition to "urge" was checked. The average daily number of UUI episodes was calculated using the daily entries in the PVD (which was to be completed prior to each study visit) as the total number of UUI episodes that occurred on a CDD divided by the number of CDDs in the PVD. CFB was calculated as the post-BL value minus the BL value. "Per 24 hours" corresponds to one Diary Day (i.e., time between when participant got up for the day each morning and time participant got up for the day the next morning as recorded in the PVD). Covariates included in the MMRM were study visit, treatment, treatment by study visit interaction, Baseline, and the statistically significant terms in Study RVT-901-3003: sex. Only participants with evaluable data were analyzed.
Time Frame: Baseline; Week 52
Population: Full Analysis Set Extension for Incontinence (FAS-Ext-I) Population: all randomized OAB Wet participants who were included in the FAS-I population in Study RVT-901-3003, who took at least 1 dose of double-blind study treatment in this extension study and had at least 1 subsequent evaluable CFB UUI measurement.
Measure: Least Squares Mean (Standard Error); unit: UUI episodes per 24 hours
Groups:
- 52 Weeks Vibegron 75 mg: Participants who met the definition of OAB Wet at study entry (based on the PVD and had been randomized in Study RVT-901-3003 to receive vibegron 75 milligrams (mg) were to continue their same treatment once daily in a blinded fashion for 40 weeks. Thus, through participation in both Study RVT-901-3003 and this extension study, participants originally randomized to vibegron 75 mg were to receive 52 weeks total of vibegron. OAB Wet participants were those participants with an average of ≥8.0 micturitions per Diary Day (DD); with an average of ≥1.0 UUI episodes per DD; and, if stress urinary incontinence (SUI) was present, with a total number of UUI episodes greater than the total number of SUI episodes from the previous visit diary. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
- 52 Weeks Tolterodine ER 4 mg: Participants who met the definition of OAB Wet at study entry (based on the PVD and had been randomized in Study RVT-901-3003 to receive tolterodine ER 4 mg were to continue their same treatment once daily in a blinded fashion for 40 weeks. Thus, through participation in both Study RVT-901-3003 and this extension study, participants originally randomized to tolterodine ER 4 mg were to receive 52 weeks total of tolterodine ER. OAB Wet participants were those participants with an average of ≥8.0 micturitions per Diary Day (DD); with an average of ≥1.0 UUI episodes per DD; and, if stress urinary incontinence (SUI) was present, with a total number of UUI episodes greater than the total number of SUI episodes from the previous visit diary. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
Arm/Group | 52 Weeks Vibegron 75 mg | 52 Weeks Tolterodine ER 4 mg
Number analyzed (Participants) | 125 | 91
UUI episodes per 24 hours | -2.2 (0.15) | -1.7 (0.17)
Statistical Analysis 1: Comparison: 52 Weeks Vibegron 75 mg; Test type: Other — Estimation of within treatment group change from Baseline; Least squares mean = -2.2, 95% CI 2-sided [-2.5 to -1.9]
Statistical Analysis 2: Comparison: 52 Weeks Tolterodine ER 4 mg; Test type: Other — Estimation of within treatment group change from Baseline; Least squares mean = -1.7, 95% CI 2-sided [-2.0 to -1.3]

4. Secondary Outcome: CFB at Week 52 in the Average Number of Urgency Episodes (Need to Urinate Immediately) Over 24 Hours in All OAB Participants
Description: The number of urgency episodes is defined as the number of times a participant had checked "need to urinate immediately" on a CDD divided by the number of CDDs in the PVD. CFB is calculated as the post-BL value minus the BL value. "Over 24 hours" corresponds to one Diary Day (i.e., time between when the participant got up for the day each morning and time the participant got up for the day the next morning as recorded in the PVD). Covariates included in the MMRM were study visit, treatment, treatment by study visit interaction, Baseline, and the statistically significant terms in Study RVT-901-3003: OAB type (Wet versus Dry) and sex.
Time Frame: Baseline; Week 52
Population: FAS-Ext Population. Only participants with evaluable data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: urgency episodes over 24 hours
Arm/Group | 52 Weeks Vibegron 75 mg | 52 Weeks Tolterodine ER 4 mg
Number analyzed (Participants) | 152 | 120
urgency episodes over 24 hours | -3.4 (0.34) | -3.2 (0.37)
Statistical Analysis 1: Comparison: 52 Weeks Vibegron 75 mg; Test type: Other — Estimation of within treatment group change from Baseline; Least squares mean = -3.4, 95% CI 2-sided [-4.0 to -2.7]
Statistical Analysis 2: Comparison: 52 Weeks Tolterodine ER 4 mg; Test type: Other — Estimation of within treatment group change from Baseline; Least squares mean = -3.2, 95% CI 2-sided [-4.0 to -2.5]

5. Secondary Outcome: CFB at Week 52 in the Average Number of Total Urinary Incontinence Episodes Over 24 Hours in OAB Wet Participants
Description: The number of total incontinence episodes is defined as the number of times a participant had checked the accidental urine leakage box in the PVD, including for reasons of "urge," "stress," or "other." CFB was calculated as the post-BL value minus the BL value. "Over 24 hours" corresponds to one Diary Day (i.e., time between when the participant got up for the day each morning and time the participant got up for the day the next morning as recorded in the PVD). Covariates included in the MMRM were study visit, treatment, treatment by study visit interaction, Baseline, and the statistically significant terms in Study RVT-901-3003: sex. hr = hour.
Time Frame: Baseline; Week 52
Population: FAS-Ext-I Population. Only participants with evaluable data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Urinary incontinence episodes over 24 hr
Arm/Group | 52 Weeks Vibegron 75 mg | 52 Weeks Tolterodine ER 4 mg
Number analyzed (Participants) | 125 | 91
Urinary incontinence episodes over 24 hr | -2.5 (0.17) | -1.9 (0.19)
Statistical Analysis 1: Comparison: 52 Weeks Vibegron 75 mg; Test type: Other — Estimation of within treatment group change from Baseline; Least squares mean = -2.5, 95% CI 2-sided [-2.8 to -2.2]
Statistical Analysis 2: Comparison: 52 Weeks Tolterodine ER 4 mg; Test type: Other — Estimation of within treatment group change from Baseline; Least squares mean = -1.9, 95% CI 2-sided [-2.3 to -1.6]

ADVERSE EVENTS:
Time Frame: up to 56 weeks
Description: Treatment-emergent adverse events were collected in members of the Safety Set Extension, comprised of all participants who received at least one dose of double-blind study treatment during RVT-901-3004. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data.
Arm/Group | Overall Vibegron 75 mg | Overall Tolterodine ER 4 mg
All-Cause Mortality (participants affected / at risk) | 1/273 | 0/232
Serious Adverse Events (participants affected / at risk) | 9/273 | 10/232
Other Adverse Events (participants affected / at risk) | 65/273 | 56/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Vibegron 75 mg (N=273) | Overall Tolterodine ER 4 mg (N=232)
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis microscopic (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Vibegron 75 mg (N=273) | Overall Tolterodine ER 4 mg (N=232)
Dry mouth (Gastrointestinal disorders) | 5 | 12
Nasopharyngitis (Infections and infestations) | 13 | 12
Urinary tract infection (Infections and infestations) | 18 | 17
Headache (Nervous system disorders) | 15 | 9
Hypertension (Vascular disorders) | 24 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor does not object to publication by Institution or Principal Investigator (PI) of results of the Trial based on information collected or generated by the Institution or PI. However, the Institution and PI are required to provide the Sponsor with an opportunity to review any proposed publication or other type of disclosure before it is submitted or otherwise disclosed to ensure against any inadvertent disclosure of Sponsor Confidential Information or unprotected Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT03583372/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT03583372/SAP_001.pdf